CLINICAL TRIAL: NCT01713400
Title: Tacrolimus, Sirolimus and Ustekinumab vs. Tacrolimus and Sirolimus for the Prevention of Acute Graft-Versus-Host Disease Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: Tacrolimus, Sirolimus and Ustekinumab vs. Tacrolimus and Sirolimus for the Prevention of Acute Graft-Versus-Host Disease
Acronym: Ustekinumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCC-16743
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Graft vs. Host Disease
Keywords: Acute Graft vs. Host Disease (aGVHD); Graft vs. Host Disease (GVHD)
MeSH Terms: conditions — Graft vs Host Disease | interventions — Ustekinumab; Sodium Chloride; Tacrolimus; Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ustekinumab (Experimental): Ustekinumab, Tacrolimus and Sirolimus. Ustekinumab: 45 mg for adults who weight 100 kg or less; 90 mg for adults who weight greater than 100 kg. Tacrolimus: Level determined according to Blood and Marrow Transplant (BMT) Program standard operating procedures. Sirolimus: The dose for both loading and ongoing administration to be dictated by the standard operating procedures of the BMT program.
  Interventions: Drug: Ustekinumab; Drug: Tacrolimus (TAC); Drug: Sirolimus
- Placebo (Placebo Comparator): Placebo, Tacrolimus, and Sirolimus. Placebo: Identical volume to that of ustekinumab. Tacrolimus: Level determined according to Blood and Marrow Transplant (BMT) Program standard operating procedures. Sirolimus: The dose for both loading and ongoing administration to be dictated by the standard operating procedures of the BMT program.
  Interventions: Drug: Placebo; Drug: Tacrolimus (TAC); Drug: Sirolimus

INTERVENTIONS:
Drug: Ustekinumab — One subcutaneous injection administered on day -1 and repeated on day +20 after transplant
  Other Names: STELARA
  Arms: Ustekinumab
Drug: Placebo — Subcutaneous injection of sterile saline (identical volume to that of ustekinumab) administered via the identical route and schedule as ustekinumab.
  Other Names: saline
  Arms: Placebo
Drug: Tacrolimus (TAC) — Administered starting day -3 according to Blood and Marrow Transplant (BMT) Program standard operating procedures. TAC levels to be monitored and maintained at a target range of 3-7 given concurrent administration with sirolimus. Specific dose adjustments within this therapeutic range to be determined by the treating physician.
  Other Names: TAC; Protopic; Prograf; Hecoria
Drug: Sirolimus — Administered initially as an oral loading dose on day -1. Thereafter, SIR to be administered as an oral regimen daily. The dose for both loading and ongoing administration to be dictated by the standard operating procedures of the BMT program. SIR levels to be monitored according to standard procedures. Dose adjustments to be made according to drug levels, with target range of 5-14ng/mL (therapeutic range by Abbott Architect instrument at Moffitt).
  Other Names: SIR; Rapamune

SUMMARY:
To determine whether treatment with ustekinumab will alter the ratio of T Regulatory Cell (Treg)/total cluster of differentiation 4 (CD4)+ cells in peripheral blood at day 30 post-hematopoietic cell transplantation (HCT).

DETAILED DESCRIPTION:
This is a comparative study to assess the biologic and clinical activity of the agent ustekinumab when given in concert with our established regimen of SIR/TAC. Patients will be randomly assigned between the standard regimen of tacrolimus/sirolimus (TAC/SIR + placebo) vs. the investigational regimen of tacrolimus/sirolimus/ustekinumab (TAC/SIR/U) in a 1:1 scheme.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic disorder requiring allogeneic hematopoietic cell transplantation
* Adequate vital organ function:
* Left ventricular ejection fraction (LVEF) >/= 45% by multigated acquisition (MUGA) scan
* FEV1, FVC, and diffusing lung capacity oxygenation (DLCO) >/= 50% of predicted values on pulmonary function tests
* Transaminases (AST, ALT) < 3 times upper limit of normal values
* Creatinine clearance >/= 50 cc/min.
* Performance status: Karnofsky Performance Status Score >/= 60%.

Exclusion Criteria:

* Active infection not controlled with appropriate antimicrobial therapy
* HIV, hepatitis B, or hepatitis C infection
* Sorror's co-morbidity factors with total score > 3
* Important modification to co-morbidity index calculation: DLCO will not be included in assessment of pulmonary risk, excepting those with DLCO < 50%, who will merit a score of 3 and thereby be excluded from the trial.
* Anti-thymocyte globulin (ATG) as part of the conditioning regimen
* Cyclophosphamide as part of the conditioning regimens

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pidala, MD, MS, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Pidala J, Beato F, Kim J, Betts B, Jim H, Sagatys E, Levine JE, Ferrara JLM, Ozbek U, Ayala E, Davila M, Fernandez HF, Field T, Kharfan-Dabaja MA, Khaira D, Khimani F, Locke FL, Mishra A, Nieder M, Nishihori T, Perez L, Riches M, Anasetti C. In vivo IL-12/IL-23p40 neutralization blocks Th1/Th17 response after allogeneic hematopoietic cell transplantation. Haematologica. 2018 Mar;103(3):531-539. doi: 10.3324/haematol.2017.171199. Epub 2017 Dec 14. PMID 29242294
- See also: H. Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 participants (potential donors and recipients) were enrolled at Moffitt Cancer Center from 3/15/2013 through 5/22/2014.
Pre-assignment Details: 30 eligible recipients were randomly assigned 1:1 (Ustekinumab n=15, Placebo n=15) with stratification for donor type. Results Data pertains to recipients only.
Period: Overall Study
Arm/Group | Ustekinumab | Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participating recipients
Groups:
- Total: Total of all reporting groups
Arm/Group | Ustekinumab | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: T Regulatory Cell (Treg)/Total Cluster of Differentiation 4 (CD4)+ Ratio
Description: Median Blood Treg/Total CD4+ Ratio at day 30 following hematopoietic cell transplantation (HCT). Comparison between study arms: Ustekinumab vs. Placebo. From NCI Dictionary: "T reg" - A type of immune cell that blocks the actions of some other types of lymphocytes, to keep the immune system from becoming over-active. T regs are being studied in the treatment of cancer. A T reg is a type of white blood cell and a type of lymphocyte. Also called regulatory T cell, suppressor T cell, and T-regulatory cell.
Time Frame: 30 days post transplant
Population: All participating recipients
Measure: Median (Full Range); unit: ratio
Arm/Group | Ustekinumab | Placebo
Number analyzed (Participants) | 15 | 15
ratio | 13 [2 to 22] | 11 [3 to 20]

2. Secondary Outcome: Incidence of Acute Graft vs. Host Disease (AGVHD)
Description: Cumulative incidence of Grade II - IV AGVHD to be characterized weekly from day of transplant to day 100 using the 1995 updated grading scheme for Graft vs. Host Disease (GVHD) developed by Glucksberg, et al.
Time Frame: 100 days post transplant
Population: All participating recipients
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab | Placebo
Number analyzed (Participants) | 15 | 15
percentage of participants | 33.3 | 40.0

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | Ustekinumab | Placebo
Serious Adverse Events (participants affected / at risk) | 4/15 | 4/15
Other Adverse Events (participants affected / at risk) | 8/15 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab (N=15) | Placebo (N=15)
Blood and lymphatic system disorders - Other, TMA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Acute cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, GVHD of gut (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, VOD (Hepatobiliary disorders) | 2 (2) | 1 (2)
Portal hypertension (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, HHV6 infection affecting CNS (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, renal failure-dialysis (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, GVHD of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab (N=15) | Placebo (N=15)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 2 (2) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (5) | 2 (8)
Diarrhea (Gastrointestinal disorders) | 1 (6) | 2 (2)
Rhinitis infective (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory infection (Infections and infestations) | 1 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 2 (7)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood and lymphatic disorders - Other (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (6) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (6)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 1 (5)
Blood bilirubin increased (Investigations) | 1 (3) | 0 (0)
GGT increased (Investigations) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes